CLINICAL TRIAL: NCT00608790
Title: Diagnostic Yield of Induced Sputum for Rapid Diagnosis of Pulmonary Tuberculosis
Brief Title: Rapid Diagnosis of Pulmonary Tuberculosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mark Hatherill, Associate Professor, University of Cape Town
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-0058; 5R01AI075603-04 (NIH)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, TB, Mycobacterium tuberculosis, children, South Africa
MeSH Terms: conditions — Tuberculosis | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Salbutamol; Drug: Sodium chloride 5%

INTERVENTIONS:
Drug: Salbutamol — Prophylactic salbutamol administered at a dose of 200 micrograms by metered dose inhaler (MDI) via a spacer.
Drug: Sodium chloride 5% — 30 ml sterile hypertonic saline solution (sodium chloride 5%) will be administered by jet nebulisation for 15-20 minutes.

SUMMARY:
The purpose of this study is to test whether a saline nebulization (breathing in a mist of moist air through a mask) will help an individual cough up a better sputum sample to test for tuberculosis (TB). In addition, this study will test whether samples obtained with saline nebulization are better at finding TB in people with HIV infection. The study will enroll up to 600 individuals, aged 12 and older, with suspected pulmonary TB. Participants will be asked to cough up a sample of sputum into a container. Then, participants will be asked to breathe a mist of moist air from an oxygen mask followed by moist salty air, which will help individuals to cough up a second sputum sample. This mist of moist air will contain salbutamol, a medicine to help open up the airways. The sputum samples will be sent to a laboratory to test for TB. Additionally, participants will be tested for HIV with a blood sample collection. Participants will be involved in study related procedures for up to 61 days.

DETAILED DESCRIPTION:
Early case detection, treatment, and prompt household contact investigation, depend on rapid microbiological confirmation, by direct smear microscopy of acid-fast bacilli, in patients with suspected pulmonary tuberculosis. Since delayed diagnosis may result in death due to lack of appropriate therapy, rapid microbiological diagnosis is especially critical in HIV-infected persons. Improved rapid diagnostic methods are also crucial for the success of epidemiological studies; trials of preventative interventions, such as novel vaccines; and therapeutic interventions, since the diagnostic endpoints of such trials may require microbiological confirmation of tuberculosis. In clinical practice, early therapeutic intervention might reduce the risk of death, especially in patients co-infected with HIV. In this study, researchers propose to test a simple diagnostic modality for rapid diagnosis of pulmonary tuberculosis in HIV-infected and HIV-uninfected adolescents and adults. Researchers will test whether induced sputum will improve the diagnostic yield of smear positive tuberculosis. This low-cost technology augments spontaneous sputum production by inhalation of a nebulized saline solution. The primary objective of this study is to quantify and compare the diagnostic yield of smear positive tuberculosis from induced sputum, with that of routine sputum, in HIV-infected patients with suspected tuberculosis. Researchers believe that induced sputum will increase the diagnostic yield from direct smear microscopy in this patient population. The secondary objective of the study is to quantify and compare the diagnostic yield of smear positive tuberculosis from induced sputum, with that of routine sputum, in all patients with suspected tuberculosis, regardless of HIV status. Researchers believe that induced sputum will increase the diagnostic yield from direct smear microscopy in all patients in this population, regardless of HIV status. Approximately 1200 individuals (male or female gender), aged 12 years and older, with suspected pulmonary tuberculosis, will be screened in order to enroll 600 eligible participants at 2 district health services clinics near the town of Worcester, Western Cape Province, South Africa. Informed consent for participation will be sought from adolescents and adults with suspected pulmonary tuberculosis who present to public sector community health services for investigation. A rapid HIV test, with pre- and post-test counseling, will be performed. A routine spontaneous expectorated sputum sample and an induced sputum sample (obtained after nebulization of sterile 5% saline via mask) will be collected. A second routine sputum will be collected on the following morning. Direct smear microscopy and mycobacterial culture of sputum will be performed in an accredited microbiology laboratory. HIV rapid test results will be used to classify participants for evaluation of the primary outcome, positive direct smear microscopy, and the secondary outcome, positive culture of M. tuberculosis. Diagnostic yields for each routine and induced sputum sample will be calculated, as a proportion of all patients who are culture-positive for M. tuberculosis, and compared in a pair-wise and sequential manner. Results will be reported as differences in yield and 95% confidence intervals for the difference in those proportions. The primary endpoint will be sputum direct smear microscopy positive for acid-fast bacilli. The secondary endpoint will be sputum culture positive for Mycobacterium tuberculosis. Study duration will be 4 years with individual subject participation approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

Adolescents and adults with suspected pulmonary tuberculosis who are referred, or self-refer, to health services clinics for investigation for tuberculosis, will be eligible to participate.

Exclusion Criteria:

* Failure to obtain informed consent (including failure to consent for either sputum collection procedures or failure to consent for HIV testing);
* Age less than 12 years;
* A history of asthma;
* A history of heart disease;
* A history of cardiac arrhythmia;
* Inability to tolerate sputum induction procedures;
* Inability to return for study follow-up visit;
* Need for hospital-based in-patient treatment or supplemental oxygen therapy;
* Other acute or chronic lung disease that may compromise lung function;
* Current anti-tuberculous therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Sputum direct smear positive for acid-fast bacilli. | Day 56 +

SECONDARY OUTCOMES:
Sputum culture positive for Mycobacterium tuberculosis. | Day 56 +

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, MD, FCPaed, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Derived] Geldenhuys HD, Whitelaw A, Tameris MD, Van As D, Luabeya KK, Mahomed H, Hussey G, Hanekom WA, Hatherill M. A controlled trial of sputum induction and routine collection methods for TB diagnosis in a South African community. Eur J Clin Microbiol Infect Dis. 2014 Dec;33(12):2259-66. doi: 10.1007/s10096-014-2198-4. Epub 2014 Jul 15. PMID 25022447